CLINICAL TRIAL: NCT00581620
Title: To Evaluate the Humoral Immune Response to a Conjugated Pneumococcus Vaccine 7-Valent (Prevenar®) in Children From High Risk Groups.
Brief Title: Study Evaluating Prevenar Immunogenicity in High Risk Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0887X-100974
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine
Keywords: pneumococcus conjugated vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- G1 (Active Comparator): G1: HIV+
  Interventions: Biological: pneumococcus conjugate vaccine
- G2 (Active Comparator): G2: Sicle Cell disease
  Interventions: Biological: pneumococcus conjugate vaccine
- G3 (Active Comparator): G3: neprotic symdrome
  Interventions: Biological: pneumococcus conjugate vaccine
- G4 (Active Comparator): G4: Chronic pulmonary disease
  Interventions: Biological: pneumococcus conjugate vaccine

INTERVENTIONS:
Biological: pneumococcus conjugate vaccine — Infants from 1 to 6 months: 3 doses at 2; 4; 6 m and booster from 12 to 15 months.

SUMMARY:
To determine immunogenicity of the heptavalent CRM197 pneumococcal conjugate in children with immunodeficiency condition. To evaluate tolerability of Prevenar® in that population.

DETAILED DESCRIPTION:
This study will require 24 months to be completed. Each child will participate for a period of time according to age of the 1st dose of vaccination: infants up to 6 months of age will be evaluated for 5 months; infants between 7 to 11 months will be evaluated for 3 months; children between 12 months up to 9 years of age will be evaluate for 2 months

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 months to 9 years old.
* Children with HIV+; Sickle Cell disease; Neprotic symdrome; Chronic pulmonary disease
* No history of seizures

Ages: 2 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2002-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine immunogenicity of the heptavalent CRM197 pneumococcal conjugate in children with immunodeficiency condition | 4 months

SECONDARY OUTCOMES:
To evaluate tolerability of Prevenar* in that population. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer